CLINICAL TRIAL: NCT00574912
Title: A Comparison of PK/PD Dose Response Characteristics of Glargine in Type 2 Diabetics
Brief Title: Characteristics of Glargine in Type 2 Diabetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Steve Davis, Chairman of Medicine, University of Maryland, Baltimore, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#060887-Lantus Glargine; VUMC 32787
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Results first posted 2015-08-03 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Insulin Glargine; Endogenous Glucose Production
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Placebo then Insulin Glargine (Experimental): Placebo: administer single dose of Placebo subcutaneously (SC) with blood glucose monitoring over 24 hours.
  Then Insulin Glargine SQ 8 weeks later, in increasing doses (0.5, 1.0, 1.5, 2.0 u/kg body wt.) with blood glucose monitoring monitoring over a 24 hour period. Each dose is separated by 8 weeks (5 separate study visits)
  Interventions: Drug: Placebo; Drug: Insulin Glargine 0.5 u/kg body wt SC; Drug: Insulin Glargine 1.0 u/kg body wt SC; Drug: Insulin Glargine 1.5 u/kg body wt SC; Drug: Insulin Glargine 2.0 u/kg body wt SC

INTERVENTIONS:
Drug: Placebo — single dose of Placebo injected s/c at 8am and monitor blood glucose over 24 hours
  Other Names: Lantus
Drug: Insulin Glargine 0.5 u/kg body wt SC — 8 weeks later, a differing dose (0.5, 1.0, 1.5, 2.0 u/kg body wt.) of Insulin Glargine and monitoring over a 24 hour period each separated by 8 weeks (5 separate study visits)
  Other Names: Lantus
Drug: Insulin Glargine 1.0 u/kg body wt SC
  Other Names: Lantus
Drug: Insulin Glargine 1.5 u/kg body wt SC
  Other Names: Lantus
Drug: Insulin Glargine 2.0 u/kg body wt SC
  Other Names: Lantus

SUMMARY:
The study is to determine the dose response relationship of insulin glargine in type 2 diabetes over a 24-hour period and measuring the differences in glucose production among the differing doses of glargine.

Hypothesis: Differing doses of insulin glargine over a 24-hour period in type 2 diabetes will show differing effects on endogenous glucose production, glucose disposal and carbohydrate and lipid flux.

DETAILED DESCRIPTION:
The incidence of type 2 DM is increasing worldwide at an alarming rate. Unfortunately, the number of individuals with glycemic control at or below the American Diabetes Association goal of 7% has dropped. In fact, the number of patients with their important cardiometabolic risk factors of glucose, lipids and blood pressure at goal is only 7%. One of the reasons for this lack of metabolic control in type 2 DM is the continued relative underutilization of insulin. Diabetes is an insulin deficient state and requires appropriate physiologic replacement of insulin. Physiologic replacement of insulin requires a basal component to restrain overnight endogenous glucose production, lipolysis and proteolysis. The other component involves prandial insulin to regulate post prandial glucose levels. Recently, insulin glargine was introduced as a once-a-day peakless basal insulin. This form of basal insulin reproduces the normal constitutive physiologic release of insulin from the pancreas. Insulin glargine represents a breakthrough in treatment as the previous available "basal insulins" either produced peaks of activity (which are disadvantageous as this results in hypoglycemia) or do not last 24 hrs which results in post absorbative hyperglycemia. Despite the undoubted advantages of insulin glargine, there remains a lack of information regarding some aspects of glargine action. The study objectives are: 1) to determine the pharmacokinetic and pharmacodynamic dose response relationship of insulin glargine in Type 2 DM; 2) partition the dose response relationship of insulin glargine on endogenous glucose production and glucose uptake in Type 2 DM; and 3) to determine if the pharmacokinetic and pharmacodynamics of insulin glargine are consistent over a wide range of doses.

ELIGIBILITY:
Inclusion Criteria:

* 12 adults (males or females) with type 2 diabetes for at least six (6) months. May be using oral agents (SUs, metformin, acarbose or glitinides) with or without insulin.
* HgbA1c 7 -12%
* Age 18-70 years
* BMI 27-40 kg/m²

Exclusion Criteria:

* Any past or present clinically relevant abnormality, medical condition, or circumstance making the subject unsuitable for participation in the study
* Evidence of hepatic, renal or cardiac failure
* Abnormal results following screening tests
* Pregnant or lactating females or females of childbearing potential who are unwilling to abstain from sexual intercourse or use reliable, medically accepted methods of contraception
* Currently using TZDs
* History of alcoholism or drug abuse within 12 months of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-03; Primary Completion 2009-09 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N. Davis, MD, FRCP, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Wang Z, Hedrington MS, Gogitidze Joy N, Briscoe VJ, Richardson MA, Younk L, Nicholson W, Tate DB, Davis SN. Dose-response effects of insulin glargine in type 2 diabetes. Diabetes Care. 2010 Jul;33(7):1555-60. doi: 10.2337/dc09-2011. Epub 2010 Mar 31. PMID 20357371

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 individuals will be their own controls completing 5 separate 24 hour protocol studies. If a participant does not complete all protocols, another person will be recruited to complete the protocols until there are 12 completed studies in each arm/group.
Groups:
- 1 All Interventions: Other: 1--All interventions
  All participant will be given all 5 interventions in the same order
  Placebo, then 0.5 units of Glargine/kg body weight, then 1.0 units of Glargine/kg body weight, then 1.5 units of Glargine/kg body weight, then 2.0 units of Glargine/kg body weight,
Period: Overall Study
Arm/Group | 1 All Interventions
Started | 20
Completed Placebo | 12 (12 original participants started the trial.)
Completed 0.5 | 12
Completed 1.0 | 12
Completed 1.5 | 12
Completed 2.0 | 12
Completed | 12
Not Completed | 8
Not completed — Could not place IV lines. | 3
Not completed — scheduling conflicts | 3
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: One participant may have received more than one intervention.
Groups:
- 1--All Interventions: Arm: Other: 1--All interventions
  All participant will be given all 5 interventions in the same order
  Placebo, then 0.5 units of Glargine/kg body weight, then 1.0 units of Glargine/kg body weight, then 1.5 units of Glargine/kg body weight, then 2.0 units of Glargine/kg body weight,
Arm/Group | 1--All Interventions
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Glucose Infusion Rate
Description: measuring the changes in glucose infusion rate during the 24 hour experimental period.
Time Frame: 24 hours
Population: 12 participants in each arm
Measure: Mean (Standard Error); unit: umol/kg/min
Groups:
- Placebo; 0.5 Units of Glargine/kg; 1.0 Units of Glargine/kg; 1.5 Units of Glargine/kg; 2.0 Units of Glargine/kg: Maximum glucose infusion rate
Arm/Group | Placebo | 0.5 Units of Glargine/kg | 1.0 Units of Glargine/kg | 1.5 Units of Glargine/kg | 2.0 Units of Glargine/kg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
umol/kg/min | 0.3 (0.3) | 2.6 (0.9) | 5.5 (1.5) | 6.8 (2.0) | 9.5 (2.1)
Statistical Analysis 1: Comparison: Placebo vs 0.5 Units of Glargine/kg vs 1.0 Units of Glargine/kg vs 1.5 Units of Glargine/kg vs 2.0 Units of Glargine/kg; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Placebo: Placebo
  Insulin Glargine: administering single, differing dose of insulin glargine over a 24 hour period every 8 weeks times five
- 0.5 Units of Glargine/kg Body Weight: 0.5 units of Glargine/kg body weight
  Insulin Glargine: administering single, differing dose of insulin glargine over a 24 hour period every 8 weeks times five
- 1 Unit of Glargine/kg Body Weight: 1 unit of glargine/kg body weight
  Insulin Glargine: administering single, differing dose of insulin glargine over a 24 hour period every 8 weeks times five
- 1.5 Units of Glargine/kg Body Weight: 1.5 units of glargine/kg body weight
  Insulin Glargine: administering single, differing dose of insulin glargine over a 24 hour period every 8 weeks times five
- 2.0 Units of Glargine/kg Body Weight: 2.0 units of glargine/kg body weight
  Insulin Glargine: administering single, differing dose of insulin glargine over a 24 hour period every 8 weeks times five
Arm/Group | Placebo | 0.5 Units of Glargine/kg Body Weight | 1 Unit of Glargine/kg Body Weight | 1.5 Units of Glargine/kg Body Weight | 2.0 Units of Glargine/kg Body Weight
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No